CLINICAL TRIAL: NCT00770588
Title: A Placebo-Controlled, Multicentre, Randomised, Parallel Group, Trial to Assess the Efficacy, Safety and Tolerability of Gefitinib (Iressa® 250mg) as Maintenance Therapy in Locally Advanced or Metastatic (StageIIIB/IV) Non Small Cell Lung Cancer (NSCLC) Chinese Patients Who HaveNot Experienced Disease Progression or Unacceptable Toxicity During Front Line Standard Platinum-Based Chemotherapy
Brief Title: Assess the Efficacy, Safety and Tolerability of Gefitinib (Iressa® 250mg) as Maintenance Therapy in Locally Advanced or Metastatic (Stage IIIB/IV) Non Small Cell Lung Cancer (NSCLC)
Acronym: INFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7913L00071; NCT00769639 (obsolete NCT alias)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2012-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer (NSCLC); Gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gefitinib (Experimental): Gefitinib (Iressa® 250 mg) 1 tablet daily
  Interventions: Drug: Gefitinib
- placebo (Placebo Comparator): placebo 1 tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefitinib — Dose form: 250 mg/tablet; Route: oral; Frequency: 1 tablet per day; Duration: until to objective PD
  Other Names: Iressa
  Arms: gefitinib
Drug: Placebo — To match Gefitinib
  Arms: placebo

SUMMARY:
This is a double blind, multicentre, randomized, placebo-controlled study. The eligible patients will be randomized to receive gefitinib or placebo at 1:1 ratio. This study will recruit 296 male or female, histologically or cytologically diagnosed locally advanced or metastatic NSCLC patients with a World Health Organization (WHO) Performance Status (PS) 0-2. Patients must have completed 4 cycles of platinum based first line doublet chemotherapy without experiencing disease progression or unacceptable toxicity. The chemotherapy shall be given every 3 weeks, which includes cisplatin or carboplatin, combined with any one of the following: gemcitabine, paclitaxel, docetaxel, vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic (stage=IIIB/IV) non-small cell lung cancer (NSCLC) before the front line chemotherapy. Note: sputum cytology alone is not acceptable
* Patients have completed 4 cycles of first line platinum contained doublet chemotherapy without progression or intolerable toxicity.
* Patients with PR or SD on study entry need to have one or more measurable lesions according to RECIST criteria.
* The study treatment should be started at least 3 weeks (21 days) but no more than 6 weeks (42 days) since last dose of chemotherapy, and within 4 weeks (28 days) since last tumour assessment.

Exclusion Criteria:

* Prior exposure to monoclonal antibodies or small molecule inhibitors against EGFR receptors. (e.g. gefitinib, erlotinib, C225)
* Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they are clinically stable and have been discontinued from steroid therapy for at least 4 weeks prior to first dose of study medication.
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* Known biomarker status of one or more of the following: Tumour EGFR gene copy number, tumour EGFR gene mutation status, tumour EGFR protein expression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shengyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhao H, Fan Y, Ma S, Song X, Han B, Cheng Y, Huang C, Yang S, Liu X, Liu Y, Lu S, Wang J, Zhang S, Zhou C, Wang M, Zhang L; INFORM investigators. Final overall survival results from a phase III, randomized, placebo-controlled, parallel-group study of gefitinib versus placebo as maintenance therapy in patients with locally advanced or metastatic non-small-cell lung cancer (INFORM; C-TONG 0804). J Thorac Oncol. 2015 Apr;10(4):655-64. doi: 10.1097/JTO.0000000000000445. PMID 25546556
- [Derived] Zhang L, Ma S, Song X, Han B, Cheng Y, Huang C, Yang S, Liu X, Liu Y, Lu S, Wang J, Zhang S, Zhou C, Zhang X, Hayashi N, Wang M; INFORM investigators. Gefitinib versus placebo as maintenance therapy in patients with locally advanced or metastatic non-small-cell lung cancer (INFORM; C-TONG 0804): a multicentre, double-blind randomised phase 3 trial. Lancet Oncol. 2012 May;13(5):466-75. doi: 10.1016/S1470-2045(12)70117-1. Epub 2012 Apr 17. PMID 22512843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 298 patients were screened for the study and 296 subsequently randomized
Period: Overall Study
Arm/Group | Gefitinib | Placebo
Started | 148 | 148
Completed | 67 | 53
Not Completed | 81 | 95
Not completed — Adverse Event | 9 | 2
Not completed — Death caused by progression of disease | 70 | 91
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefitinib | Placebo | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Customized [Number; unit: Participants]
  <45 years | 22 | 22 | 44
  45-64 years | 107 | 108 | 215
  65-74 years | 18 | 17 | 35
  >=75 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 56 | 121
  Male | 83 | 92 | 175
Smoking status [Number; unit: Participants]
  non-smoker | 79 | 81 | 160
  ex-smoker | 57 | 55 | 112
  current smoker | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS will be calculated from the tumour measurements collected at each tumour assessment per the RECIST criteria and/or the date of patient death. Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first.The primary analysis of PFS will be performed when at least 265 events have occurred, which is expected to occur approximately.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 148 | 148
month | 4.8 [3.19 to 8.54] | 2.6 [1.61 to 2.76]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS will be assessed from the time of randomisation to death from any cause. For patients not known to have died(which may include those who have been lost to follow up or who have withdrawn from the study for whatever reason), OS will be censored for the analysis at the last date at which the patients were known to be alive.
Time Frame: The OS will be assessed from the time of randomization to death from any cause.For patients not known to have died or who have withdrawn from the study for whatever reason,OS will be censored at the last date at which patients were known to be alive.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 148 | 148
month | 18.7 [15.6 to 22.2] | 16.9 [14.5 to 19.0]

3. Secondary Outcome: Objective Tumour Response (ORR)
Description: The objective tumour response will be calculated as the number of patients with CR or PR per RECIST Criteria. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: TTumour assessment using RECIST will be performed at baseline then every 42 days (6 weeks) ± 7 days (1 week) from randomisation until objective progression or death from any cause.
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 148 | 148
Participants | 35 | 1

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR will be calculated as the number of patients with CR, PR or sustained SD≥6 weeks per RECIST Criteria. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase
Time Frame: Tumour assessment using RECIST will be performed at baseline then every 42 days (6 weeks) ± 7 days (1 week) from randomisation until objective progression or death from any cause.
Reporting Status: Not Posted
Measure: Number; unit: Participants

5. Secondary Outcome: Symptom Improvement
Description: Symptom improvement will be assessed from the 7-question Lung Cancer Subscale domain score derived from the FACT-L questionnaire. It is defined as an increase of two or more points on the LCS from randomization, maintained for 21 or more days. It will be calculated as the number of patients analysed with improvement.
Time Frame: at randomization, every 6 weeks until disease progression, and at discontinuation.
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 148 | 148
Participants | 34 | 12

6. Secondary Outcome: Adverse Event
Description: Appropriate description of AEs and laboratory data/vital signs will be produced. Number of patients who had at least one adverse events will be calculated.
Time Frame: AEs and SAEs must be collected from the time that the main study informed consent is obtained to 28 days after discontinuation of study drug. Any ongoing AE or SAE at discontinuation of study treatment and during 28 day follow-up period must be monitored
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 147 | 148
Participants | 118 | 79

ADVERSE EVENTS:
Arm/Group | Gefitinib | Placebo
Serious Adverse Events (participants affected / at risk) | 10/147 | 5/148
Other Adverse Events (participants affected / at risk) | 118 | 79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=147) | Placebo (N=148)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Accidental Death (General disorders) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Gefitinib | Placebo
rash (Skin and subcutaneous tissue disorders) | 73/147 | 14/148
pruritus (Skin and subcutaneous tissue disorders) | 10/147 | 7/148
dry skin (Skin and subcutaneous tissue disorders) | 9/147 | 3/148
skin exfoliation (Skin and subcutaneous tissue disorders) | 9/147 | 0/148
diarrhoea (Gastrointestinal disorders) | 37/147 | 13/148
Alanine Aminotransferase Increased (Investigations) | 31/147 | 12/148
aspartate aminotransferase increased (Investigations) | 21/147 | 6/148
transaminases increased (Investigations) | 8/147 | 2/148
cough (Respiratory, thoracic and mediastinal disorders) | 9/147 | 20/148
serious hepatic dysfunction (Investigations) | 43/147 | 16/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to collaborate in good faith with AZ regard to contents and formation of any publication and to pay due consideration to the comments, views and opinions offered by AZ. AZ shall have a period of 30 days from receipt of the proposed final manuscript to review and may require submission be delayed in order for AZ to file patent application